CLINICAL TRIAL: NCT05374330
Title: The Use of Electroacupuncture (EA) to Affect Pain, Function and Quality of Life in Patients With End Stage Knee Osteoarthritis (KOA) on a Total Knee Arthroplasty (TKA) Waitlist
Brief Title: Electroacupuncture Treatment for Those With End Stage Knee Osteoarthritis on a Total Knee Arthroplasty Waitlist
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study withdrawn
Sponsor: University of Manitoba (Other)
Responsible Party: Principal Investigator, Janine Didyk, Principle Investigator, University of Manitoba
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H2022:100
Record Dates: First submitted 2022-04-29; First posted 2022-05-16 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2024-04

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Electroacupuncture

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Electroacupuncture (Experimental): Acupuncture needles will be inserted into the body at standardized acupuncture points. Electrical current will then be applied using 2 channels of electrical current for a total of 4 points receiving electroacupuncture
  Interventions: Other: Electroacupuncture
- Sham acupuncture (Sham Comparator): Sham Acupuncture needles will be placed at standardized acupuncture points. Sham electrical current will then be applied using 2 channels / 4 points as in the electroacupuncture group. The electrical current will not be turned on.
  Interventions: Other: Electroacupuncture
- Waitlist (No Intervention): The wait list group will be required to complete questionnaires at 4 separate time points over the 12 week study period.

INTERVENTIONS:
Other: Electroacupuncture — Acupuncture needles are inserted into the body at standardized acupuncture points. An electrical current is then applied to 4 needles through 2 channels of electrical current. The sham group receives the same protocol with sham needles and sham electrical current.
  Other Names: Electrical acupuncture
  Arms: Electroacupuncture; Sham acupuncture

SUMMARY:
A 3-armed pilot randomized controlled trial: electroacupuncture, sham acupuncture and waitlist groups.

DETAILED DESCRIPTION:
The purpose of this study is to determine the efficacy of EA as a treatment strategy in the end stage knee osteoarthritis (KOA) population waiting for total knee arthroplasty (TKA). The research objectives are to 1. To determine the efficacy of EA to provide pain relief, improve function and quality of life in the end stage KOA population who are waiting for TKA. 2. To determine if EA is superior to sham EA or waiting list groups in providing pain relief, improving function and quality of life in the end stage KOA population who are waiting for TKA.

Outcome measures will be collected from all 3 groups at baseline, mid point, completion and 6 week follow up.

Participants will be recruited from the Concordia Joint Replacement Group in Winnipeg, Manitoba.

Inclusion Criteria: participants are on a waiting list for TKA and do not have a surgical date within 3 months from the start of the study.Waiting list will be defined as having had consultation with an orthopaedic surgeon and having accepted an offer a TKA. The participants will be a minimum of 45 years old and have a NPRS ≥ 5.

Exclusion Criteria: knee pain caused by other disease or injury, arthroscopy within the past year, intra articular injection within the previous 3 months, painful ipsilateral hip OA. Participants scheduled for simultaneous bilateral TKA or revision will be excluded.

Medical history: serious acute or chronic disease or psychiatric disorders, blood coagulation disorders.

Surgical history: implanted cardiac pacemakers, history of valve replacement, previous arthroplasty.

Other: allergy to needle components, needle phobia, pregnancy

ELIGIBILITY:
Inclusion Criteria:

* participants are on a waiting list for TKA and do not have a surgical date within 3 months from the start of the study.Waiting list will be defined as having had consultation with an orthopaedic surgeon and having accepted an offer a TKA. The participants will be a minimum of 45 years old and have a NPRS ≥ 5.

Exclusion Criteria:

* Criteria: knee pain caused by other disease or injury, arthroscopy within the past year, intra articular injection within the previous 3 months, painful ipsilateral hip OA. Participants scheduled for simultaneous bilateral TKA or revision will be excluded.

Medical history: serious acute or chronic disease or psychiatric disorders, blood coagulation disorders.

Surgical history: implanted cardiac pacemakers, history of valve replacement, previous arthroplasty.

Other: allergy to needle components, needle phobia, pregnancy

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-09 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
The Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) | Baseline, 3 weeks, 6 weeks and 6 weeks after study completion
  Disease specific outcome measure. Measuring change in disease specific function over 4 time points (as noted below). The WOMAC provides a multidimensional assessment inclusive of activities of daily life (ADL's), functional mobility, gait, general health, and quality of life organized into 3 subscales (pain, stiffness, physical function) consisting of 24 items scored on a 5-point scale from 0-4. Higher scores represent higher pain values or worse function for a total possible score of 96.

SECONDARY OUTCOMES:
The Short Form-Survey 36 (SF-36) | Baseline, 3 weeks, 6 weeks and 6 weeks after study completion
  Quality of life outcome measure. Measuring change in health related QOL over 4 time points (as noted below). The SF-36 includes 36 items which cover 8 health domains: limitations in physical activities because of health problems, limitations in social activities because of physical or emotional problems, limitations in usual role activities because of physical health problems, bodily pain, general mental health, limitations in usual role activities because of emotional problems, vitality, and general health perceptions. A total score can be used to indicate low or high HRQoL, while the physical component summary and the mental component summary can be used to rate these 2 separate dimensions of HRQoL.
The Short Form McGill Pain Questionnaire (SF-MPQ) | Baseline, 2 weeks, 6 weeks, and 6 weeks after study completion
  Pain outcome measure. measuring change in pain over 4 time points (as noted below). Using a 5-point pain intensity scale, there are 4 subscales with a total of 78 pain descriptor items and a single item pain intensity scale.
Numeric Pain Rating Scale (NPRS) | Baseline, 3 weeks, 6 weeks and 6 weeks after study completion
  Pain outcome measure: measuring change in pain over 4 time points (as noted below). The NPRS measures pain on a 0-10 point scale with 0 being no pain and 10 being the most severe pain.

OTHER OUTCOMES:
Brief questionnaire | Baseline, 3 weeks, 6 weeks and 6 weeks after study completion
  asks specific questions re: pain over the course of the study, use of medication.
  and blinding. Pain is asked in a descriptive format on a 7 point scale (much better/better/slightly better/no change/slightly worse/worse/worst). Medication use is asked on 5 point scale with the use of 0-same amount, 1- much less than usual, 2- somewhat less than usual, 3- somewhat more than usual, 4-significantly less than usual. Blinding questions is asked of the electroacupuncture and sham groups "I believe that I am receiving A= True acupuncture B= Sham acupuncture

CONTACTS AND LOCATIONS:
Locations (1):
- University of Manitoba, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: No
Undetermined at this time